CLINICAL TRIAL: NCT06004596
Title: Establishing a Pediatric Reference Range for the 13C-Spirulina Gastric Emptying Breath Test (GEBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairn Diagnostics (Industry)
Collaborators: Medical College of Wisconsin (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDX-CD-PRO-442
Record Dates: First submitted 2023-05-01; First posted 2023-08-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Reference Range determination (Other): 13C-Spirulina Gastric Emptying Breath Test (GEBT) administered to healthy participants
  Interventions: Diagnostic Test: 13C-Spirulina Gastric Emptying Breath Test (GEBT)
- Biological Variability (Active Comparator): 13C-Spirulina GEBT administered a second time to subset of participants to determine pediatric biological variability.
  Interventions: Diagnostic Test: 13C-Spirulina Gastric Emptying Breath Test (GEBT); Diagnostic Test: 13C-Spirulina Gastric Emptying Breath Test (GEBT) - repeat

INTERVENTIONS:
Diagnostic Test: 13C-Spirulina Gastric Emptying Breath Test (GEBT) — Diagnostic test
Diagnostic Test: 13C-Spirulina Gastric Emptying Breath Test (GEBT) - repeat — Diagnostic test - repeat for biological variability deterination
  Arms: Biological Variability

SUMMARY:
The goal of this clinical trial is to define the normal response to the 13C-Spirulina Gastric Emptying Breath Test (GEBT) in children, so that we can use this test to help diagnose children that are suspected of having a condition called gastroparesis, which means that food doesn't empty from their stomach normally.

Participants will blow into test tubes to collect breath samples before and after eating a scrambled egg GEBT meal that contains a small amount of specially grown Spirulina (a blue-green alga used as a dietary supplement) that contains mostly carbon-13 (a non-radioactive kind of carbon atom). Analysis of the amount of 13C in the carbon dioxide in breath before and after eating the GEBT meal can measure how fast food is emptying from the stomach.

DETAILED DESCRIPTION:
Children will complete questionnaires to ensure that they are qualified to enter the study and are likely to have normal gastric emptying rates. Informed consent/assent will be obtained.

Breath samples will be collected by children blowing into test tubes before and after eating a 13C-Spirulina GEBT meal. Breath samples will be collected and the test will be administered via telehealth or at one of the children's hospital clinics.

Researchers will analyze results from different age groups to see if there are differences in normal gastric emptying in younger/older children and boys/girls.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7 to 18 years who provide written assent and whose parents provide written consent for participation
* Healthy and without any significant prior medical history or developmental delays
* Able to eat the test meal and provide breath samples.-

Exclusion Criteria:

Any known physician-diagnosed medical (gastrointestinal, pancreatic, or liver disease that may cause malabsorption, neurological) or psychiatric disease

* Chronic pulmonary disease including moderate/severe reactive airway disease requiring treatment with a daily inhaler
* Type 1 or 2 Diabetes
* Chronic gastrointestinal symptoms or functional gastrointestinal disorders
* Mental retardation or pervasive developmental disorder
* Currently receiving prescription drug therapy that may affect gastric motor function or sensation
* Any over-the-counter or herbal supplements that may affect gastric motor function or sensation
* Allergy to Spirulina, egg, milk, wheat or gluten (unless consuming gluten free crackers with the test meal) or known intolerance to any ingredient in the test meal

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
kPCD (kPCD = 1000 x percent dose of 13C excreted) at 15 minutes (min-1) | 15 minutes
  13CO2 excretion rate calculated at 15 minutes after meal completion
kPCD at 30 minutes (min-1) | 30 minutes
  13CO2 excretion rate calculated at 30 minutes after meal completion
kPCD at 45 minutes (min-1) | 45 minutes
  13CO2 excretion rate calculated at 45 minutes after meal completion
kPCD at 60 minutes (min-1) | 60 minutes
  13CO2 excretion rate calculated at 60 minutes after meal completion
kPCD at 90 minutes (min-1) | 90 minutes
  13CO2 excretion rate calculated at 90 minutes after meal completion
kPCD at 120 minutes (min-1) | 120 minutes
  13CO2 excretion rate calculated at 120 minutes after meal completion
kPCD at 150 minutes (min-1) | 150 minutes
  13CO2 excretion rate calculated at 150 minutes after meal completion
kPCD at 180 minutes (min-1) | 180 minutes
  13CO2 excretion rate calculated at 180 minutes after meal completion
kPCD at 210 minutes | 210 minutes
  13CO2 excretion rate calculated at 210 minutes after meal completion
kPCD at 240 minutes (min-1) | 240 minutes
  13CO2 excretion rate calculated at 240 minutes after meal completion
Test meal/test completion | up to 20 minutes
  Participant was able to successfully consume the meal/complete the test - Measured by determining whether box on test request form checked or not checked and whether or not all breath samples were collected/able to be analyzed
Tmax (mins) | 90 to 240 minutes
  Time of maximum excretion rate - time at which the largest kPCD is observed

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Williams, PhD, Principal Investigator — Cairn Diagnostics
Locations (3):
- United States (3):
  - Cairn Diagnostics, Brentwood, Tennessee
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No